CLINICAL TRIAL: NCT04847063
Title: Individualized Response Assessment to Heated Intraperitoneal Chemotherapy (HIPEC) for the Treatment of Peritoneal Carcinomatosis From Ovarian, Colorectal, Appendiceal, or Peritoneal Mesothelioma Histologies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 210012; 21-C-0012
Record Dates: First submitted 2021-04-14; First posted 2021-04-15 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-09-17

CONDITIONS: Peritoneal Carcinomatosis; Peritoneal Mesothelioma; Ovarian Cancer; Gastrointestinal Cancer; Appendiceal Cancer
Keywords: cytoreductive surgery (CRS); SMART System; necrosis; Ki-67; Peritoneal Metastasis
MeSH Terms: conditions — Peritoneal Neoplasms; Ovarian Neoplasms; Gastrointestinal Neoplasms; Appendiceal Neoplasms; Necrosis | interventions — Mitomycin; Cisplatin; Doxorubicin; Oxaliplatin; Fluorouracil; sodium thiosulfate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 1/ HIPEC: Oxaliplatin Randomized treatment assignment (Experimental): HIPEC with intraperitoneal oxaliplatin and IV 5-FU, randomly assigned
  Interventions: Procedure: Heated Intraperitonial Chemotherapy; Drug: Oxaliplatin; Drug: 5-Fluorouracil
- 2/ HIPEC: Mitomycin C Randomized treatment assignment (Experimental): HIPEC with intraperitoneal mitomycin C, randomly assigned
  Interventions: Drug: Mitomycin C; Procedure: Heated Intraperitonial Chemotherapy
- 3/ HIPEC: Cisplatin, Doxorubicin Randomized treatment assignme (Experimental): HIPEC with intraperitoneal cisplatin and doxorubicin, in addition to IV sodium thiosulfate, randomly assigned
  Interventions: Drug: Cisplatin; Procedure: Heated Intraperitonial Chemotherapy; Drug: Doxorubicin; Drug: Sodium Thiosulfate
- 4/ HIPEC: Cisplatin, Mitomycin C Randomized treatment assignme (Experimental): HIPEC with intraperitoneal cisplatin and mitomycin C, in addition to IV sodium thiosulfate, randomly assigned
  Interventions: Drug: Mitomycin C; Drug: Cisplatin; Procedure: Heated Intraperitonial Chemotherapy; Drug: Sodium Thiosulfate

INTERVENTIONS:
Drug: Mitomycin C — Arm 2, intraperitoneal (IP) Mitomycin C monotherapy: dosing divided into two 60-mL syringes, 30 mg per syringe. 30 mg will be given at time = 0, and the remaining 10 mg of the dose will be given at time = 60 minutes. Part of Arm 4: Mitomycin C co-therapy 15 mg/m2 for 60 minutes, given at time = 0 with cisplatin
  Arms: 2/ HIPEC: Mitomycin C Randomized treatment assignment; 4/ HIPEC: Cisplatin, Mitomycin C Randomized treatment assignme
Drug: Cisplatin — Part of Arms 3 and 4, intraperitoneal (IP)cisplatin co-therapy: 75 mg/m2 for 60 minutes, mixed in 1 L of 0.9% sodium chloride. For cisplatin-based HIPEC, intravenous sodium thiosulfate given as a loading dose of 7.5 g/m2 in 150 mL 0.9% sodium chloride at the time of introducing cisplatin into the perfusion circuit, followed by a 12-hour pump-based infusion of 25.56 g/m2 in 1 L 0.9% sodium chloride
  Arms: 3/ HIPEC: Cisplatin, Doxorubicin Randomized treatment assignme; 4/ HIPEC: Cisplatin, Mitomycin C Randomized treatment assignme
Procedure: Heated Intraperitonial Chemotherapy — Heated Intraperitonial Chemotherapy (HIPEC) with with standardized doses of chemotherapeutic agents as indicated by the subject's Arm assignment
Drug: Doxorubicin — Part of Arm 3: intraperitoneal (IP) Doxorubicin co-therapy 15 mg/m2 for 60 minutes, given at time = 0 with cisplatin
  Arms: 3/ HIPEC: Cisplatin, Doxorubicin Randomized treatment assignme
Drug: Oxaliplatin — Arm 1, intraperitoneal (IP) Oxaliplatin: 200 mg/m2 for 90 minutes, mixed in 250 mL of 5% dextrose solution. For oxaliplatin-based HIPEC, intravenous 5-fluorouracil given at a dose of 400 mg/m2 in 250 mL 0.9% sodium chloride over 10 minutes, co-administered with intravenous leucovorin at 20 mg/m2 in a separate bag of 250 mL 0.9% sodium chloride
  Arms: 1/ HIPEC: Oxaliplatin Randomized treatment assignment
Drug: 5-Fluorouracil — Part of Arm 1, for oxaliplatin-based HIPEC: intravenous 5-fluorouracil given at a dose of 400 mg/m2 in 250 mL 0.9% sodium chloride over 10 minutes, co-administered with intravenous leucovorin at 20 mg/m2 in a separate bag of 250 mL 0.9% sodium chloride
  Arms: 1/ HIPEC: Oxaliplatin Randomized treatment assignment
Drug: Sodium Thiosulfate — Part of Arms 3 and 4, for cisplatin-based HIPEC: intravenous sodium thiosulfate given as a loading dose of 7.5 g/m2 in 150 mL 0.9% sodium chloride at the time of introducing cisplatin into the perfusion circuit, followed by a 12-hour pump-based infusion of 25.56 g/m2 in 1 L 0.9% sodium chloride
  Arms: 3/ HIPEC: Cisplatin, Doxorubicin Randomized treatment assignme; 4/ HIPEC: Cisplatin, Mitomycin C Randomized treatment assignme

SUMMARY:
Background:

Cytoreductive surgery (CRS) removes tumors in the abdomen. HIPEC is heated chemotherapy that washes the abdomen. CRS and HIPEC may help people with peritoneal carcinomatosis. These are tumors that have spread to the lining of the abdomen from other cancers. Researchers think they can improve results of CRS and HIPEC by choosing the chemotherapy drugs used in HIPEC.

Objective:

To see if HIPEC after CRS can be improved, by testing different chemotherapy drugs, using a model called the SMART (Sample Microenvironment of Resected Metastatic Tumor) System.

Eligibility:

Adults ages 18 and older who have peritoneal carcinomatosis that cannot be fully removed safely with surgery.

Design:

Participants will be screened with:

Medical history

Physical exam

Blood and urine tests

Computed tomography (CAT) scan

Other imaging scans, as needed

Electrocardiogram (EKG)

Tumor biopsy, if needed

Laparoscopy. Small cuts will be made in the abdomen. A tube with a light and a camera will be used to see their organs.

Some screening tests will be repeated in the study.

Participants will enroll in NIH protocol #13C0176. This allows their tumor samples to be used in future research.

Participants will have CRS. As many of their visible tumors will be removed as possible. They will also have HIPEC. Two thin tubes will be put in their abdomen. They will get chemotherapy through one tube. It will be drained out through the other tube. They will be in the hospital for 7-21 days after surgery.

Participants will give tumor, blood, and fluid samples for research. They will complete surveys about their health and quality of life.

Participants will have follow-up visits over 5 years.

DETAILED DESCRIPTION:
Background:

Peritoneal carcinomatosis is uniformly fatal if untreated; improved outcomes are seen with aggressive cytoreductive surgery (CRS) and heated intraperitoneal chemotherapy (HIPEC).

The selection of chemotherapeutic agent for HIPEC is largely based on primary tumor histology and provider preference as opposed to knowledge of the potential efficacy of a specific agent for an individual patient.

HIPEC is intended to target small or microscopic residual disease following complete cytoreduction; however, the actual efficacy and additional benefit of HIPEC is in question.

The SMART System provides an ideal platform upon which to perfuse small peritoneal tumor tissue implants and simulate HIPEC treatment ex vivo.

Tissue response to simulated ex vivo HIPEC treatment in the SMART System could inform chemotherapeutic agent selection for subsequent cytoreduction and intra-operative in vivo HIPEC treatments.

Objective:

To determine the correlation between ex vivo simulated HIPEC in the SMART System and in vivo HIPEC with respect to two measures of response to treatment: percent necrosis and Ki-67

Eligibility:

Histologically confirmed peritoneal carcinomatosis from appendiceal, colorectal, ovarian, or peritoneal mesothelioma histologies

Absence of extra-abdominal metastatic disease

Participant deemed able to undergo complete cytoreduction

Age >= 18 years of age

Design:

This is a Phase I study of cytoreductive surgery (CRS) and heated intraperitoneal chemotherapy (HIPEC), with randomization to one of two accepted HIPEC treatment regimens as determined by primary histology.

At the time of cytoreduction, representative peritoneal tumor biopsies will be obtained before and after intra-operative in vivo HIPEC treatment.

Tumor nodules harvested before intra-operative HIPEC will be placed in the SMART System, exposed to simulated ex vivo HIPEC treatment, and then perfused, with subsequent assessment of percent necrosis and Ki-67.

Tumor nodules harvested immediately after intra-operative HIPEC will be placed in the SMART System and perfused, with subsequent assessment of percent necrosis and Ki-67.

The correlation of percent necrosis and Ki-67 assessment following simulated ex vivo HIPEC and intra-operative in vivo HIPEC will be determined.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Confirmation of peritoneal carcinomatosis from appendiceal, colorectal, ovarian, or peritoneal mesothelioma histologies by the Laboratory of Pathology, NCI.
* Measurable or evaluable disease as defined by RECIST v1.1. criteria and/or by peritoneal carcinomatosis index (PCI) score.
* Participants must be assessed to be able to undergo complete cytoreduction, with laparoscopically assessed PCI score thresholds as indicated below:

  * Primary Histology: Appendiceal/Colorectal/Ovarian / PCI Cutoff for Eligibility: Total Score < 20 (out of 39 possible points)
  * Primary Histology: Mesothelioma / PCI Cutoff for Eligibility: Total Score <= 30 (out of 39 possible points)
* Age >= 18 years.
* ECOG performance status <= 1 (Karnofsky >= 80%).
* Participants must have adequate organ and marrow function as defined below:

  * Absolute neutrophil count >= 1,000/mcL
  * Platelets >= 75,000/mcL
  * Total bilirubin within normal institutional limits
  * AST (SGOT)/ ALT (SGPT) <= 3x institutional upper limit of normal (ULN), or <= 5.0x ULN in participants with liver metastases (only)
  * Creatinine within normal institutional limits

OR

--Creatinine clearance >= 60 mL/min/1.73 m^2 for participants with creatinine levels above institutional normal calculated using eGFR.

* Because therapeutic agents used in this trial are known to be teratogenic, individuals of child-bearing potential (IOCBP) and individuals who are able to father a child must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for 180 days after last study treatment.
* Ability of participant to understand and the willingness to sign a written informed consent document.
* Ability and willingness to co-enroll on the tissue collection protocol 13C0176, Tumor, Normal Tissue and Specimens from Patients Undergoing Evaluation or Surgical Resection of Solid Tumors .

EXCLUSION CRITERIA:

* Participants with known extra-abdominal metastatic disease from the participant s appendiceal, colorectal, ovarian, or peritoneal mesothelioma primary.
* Participants who have received intraperitoneal chemotherapy or other anti-cancer therapy within the last 4 weeks prior to the start of study treatment.
* Participants who have undergone major surgery within the last 12 weeks prior to the start of study treatment.
* History of allergic reactions attributed to platinum-containing compounds.
* History of dihydropyrimidine dehydrogenase deficiency (only participants with appendiceal or colorectal cancer).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant individuals are excluded from this study because the protocol involves major abdominal surgery and chemotherapeutic agents with the potential for teratogenic or abortifacient effects. Note: Due to an unknown but potential risk for adverse events in nursing infants secondary to treatment of the participant, nursing (including breastfeeding) should be discontinued if the participant is undergoing treatment (i.e., nursing participants must agree to discontinue nursing activities).
* HIV-positive participants with detectable viral load despite antiretroviral therapy are ineligible because of participants increased risk of lethal infections when treated with marrow-suppressive therapy. HIV-positive participants who have undetectable viral load on antiretroviral therapy may be considered for this study only after consultation with a NIAID physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-10-19 (Actual); Primary Completion 2030-12-30 (Estimated); Study Completion 2031-12-30 (Estimated)

PRIMARY OUTCOMES:
To determine the correlation between ex vivo simulated HIPEC in the SMART system and in vivo HIPEC with respect to two measures of response to treatment: percent necrosis and Ki-67 | approx. 4 days post-HIPEC
  percent necrosis and Ki-67 scores will be obtained and used to determine the correlation between each measure by ex vivo simulated HIPEC in the SMART System and by in vivo intra-operative HIPEC

SECONDARY OUTCOMES:
To determine the correlation between ex vivo simulated HIPEC in the SMART System and in vivo HIPEC with respect to two measures of response to treatment: percent necrosis and Ki-67, separately within each cohort and arm subset, as well as within... | approx. 4 days post-HIPEC
  Tumor tissue responses to ex vivo simulated HIPEC and in vivo HIPEC regimens will be assessed by an intramural pathologist using percent tissue necrosis and Ki-67 scoring, both to the nearest 10 percent. These assessments will be incorporated into pathology reports following cytoreductive surgery with HIPEC
To estimate the peritoneal progression-free survival probability, separately by arms and by cohorts, in a preliminary fashion | baseline, every 3 months post-treatment for 2 years, than every 6 months for a total of 5 years
  median amount of time participant survives from time of cytoreduction until peritoneal progression, assessed for the individual cohorts and treatment arms and also compared between arms within cohorts
To estimate the peritoneal progression-free survival probability as a function of tissue response to ex vivo simulated HIPEC in the SMART System and in vivo HIPEC, as assessed by percent necrosis and Ki-67, in a preliminary fashion | baseline, every 3 months post-treatment for 2 years, than every 6 months for a total of 5 years
  median amount of time participant survives from time of cytoreduction until peritoneal progression, as assessed in tissue response by percent necrosis and Ki-67
To evaluate overall survival for up to 5 years after CRS and HIPEC | death or 5 years post-treatment
  median amount of time participant survives from CRS and HIPEC until death or for up to 5 years post-treatment
To measure Quality of Life by FACT-C and EQ-5D-5L | baseline, every 3 months post-treatment for 2 years, than every 6 months for a total of 5 years
  outcomes from QOL will be reported using descriptive statistics, as well as comparing the results from before to after treatment: physical and mental health-related quality of life, social and emotional wellbeing, and disease-related symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Blakely, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2021-C-0012.html